CLINICAL TRIAL: NCT03217266
Title: A Phase Ib Trial of Neoadjuvant AMG 232 (KRT-232) Concurrent With Preoperative Radiotherapy in Wild-Type P53 Soft Tissue Sarcoma (STS)
Brief Title: Navtemadlin and Radiation Therapy in Treating Patients With Soft Tissue Sarcoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2017-01234; NCI-2017-01234 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-DT001 (Other: NRG Oncology); NRG-DT001 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2017-07-13; First posted 2017-07-14 (Actual); Results first posted 2024-11-08 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Resectable Soft Tissue Sarcoma; Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — navtemadlin; 2-((3R,5R,6S)-5-(3-chlorophenyl)-6-(4-chlorophenyl)-1-((S)-1-(isopropylsulfonyl)-3-methylbutan-2-yl)-3-methyl-2-oxopiperidin-3-yl)acetic acid; 2-(5-(3-chlorophenyl)-6-(4-chlorophenyl)-1-(1-(isopropylsulfonyl)-3-methylbutan-2-yl)-3-methyl-2-oxopiperidin-3-yl)acetic acid; Radiotherapy; Radiation; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Step 1 (tumor tissue testing, navtemadlin) (Experimental): Patients undergo tumor tissue testing for p53 gene status and receive navtemadlin PO on days 2-4, days 2-5, or days 1-5 of weeks 1 to 5 in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Navtemadlin; Radiation: Radiation Therapy
- Step 2, Group I (navtemadlin, radiation therapy, surgery) (Experimental): Starting with week 2, patients receive navtemadlin as in Step 1 and undergo RT daily for 5 weeks in the absence of disease progression or unacceptable toxicity, followed by surgery 5-8 weeks after RT completion.
  Interventions: Drug: Navtemadlin; Radiation: Radiation Therapy; Procedure: Surgical Procedure
- Step 2, Group II (radiation therapy, surgery) (Experimental): Starting with week 2, patients undergo radiation therapy daily for 5 weeks in the absence of disease progression or unacceptable toxicity, followed by surgery 5-8 weeks after RT completion.
  Interventions: Radiation: Radiation Therapy; Procedure: Surgical Procedure

INTERVENTIONS:
Drug: Navtemadlin — Given PO
  Other Names: (3R,5R,6S)-5-(3-Chlorophenyl)-6-(4-chlorophenyl)-3-methyl-1-((1S)-2-methyl-1-(((1-methylethyl)sulfonyl)methyl)propyl)-2-oxo-3-piperidineacetic Acid; AMG 232; AMG-232; KRT 232; KRT-232; KRT232; MDM2 Inhibitor KRT-232
  Arms: Step 1 (tumor tissue testing, navtemadlin); Step 2, Group I (navtemadlin, radiation therapy, surgery)
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
Procedure: Surgical Procedure — Undergo surgery
  Other Names: Operation; Surgery; Surgery Type; Surgery, NOS; Surgical; Surgical Intervention; Surgical Interventions; Surgical Procedures; Type of Surgery
  Arms: Step 2, Group I (navtemadlin, radiation therapy, surgery); Step 2, Group II (radiation therapy, surgery)

SUMMARY:
This phase Ib trial studies the side effects of navtemadlin and radiation therapy in treating patients with soft tissue sarcoma. Navtemadlin may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Radiation therapy uses high energy x-rays to kill tumor cells and shrink tumors. Giving navtemadlin and radiation therapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety and tolerability of navtemadlin (AMG-232 [KRT-232]) in combination with standard-dose radiotherapy in soft tissue sarcoma (STS) in two separate patient cohorts (A, extremity or body wall; B, abdomen/pelvis/retroperitoneum).

II. To determine the maximum tolerated dose/recommended phase II dose (maximum tolerated dose/recommended phase 2 dosage [MTD/RP2D]) of AMG 232 (KRT-232) in combination with radiotherapy.

SECONDARY OBJECTIVES:

I. To observe and record anti-tumor activity. II. To determine percentage (%) necrosis and pathologic complete response (pCR) in final surgical resection specimen.

III. To determine % local failure (LF), disease free survival (DFS) and overall survival (OS) at 2 years.

IV. To determine pharmacodynamics (PD) effects of AMG 232 (KRT-232) when combined with radiotherapy by assessing serial serum macrophage inhibitory cytokine (MIC)-1 levels.

V. To determine AMG 232 (KRT-232) exposure (pharmacokinetics)-response relationships (PD, toxicity, and efficacy).

EXPLORATORY OBJECTIVES:

I. To determine tumor volume changes determined by magnetic resonance imaging (MRI) or computed tomography (CT) with and without contrast pre- and post-radiotherapy.

II. To characterize clinical outcomes in patients treated with AMG 232 (KRT-232) by genomic biomarkers.

III. To determine the correlation between mdm2/4 expression determined by next-generation sequencing (NGS) and the protein levels by immunohistochemistry (IHC).

IV. To explore the possibility of identifying tumor genetic mutations in (1) cell-free (cf) circulating tumor deoxyribonucleic acid (ctDNA), (2) deoxyribonucleic acid/ribonucleic acid (DNA/RNA) isolated from exosomes, and determine the concordance of these results and that from NGS.

OUTLINE: This is a dose-escalation study of navtemadlin.

STEP 1: Patients undergo tumor tissue testing for p53 gene status and receive navtemadlin orally (PO) on days 2-4, days 2-5, or days 1-5 of weeks 1 to 5 in the absence of disease progression or unacceptable toxicity.

STEP 2: Patients with a wild-type p53 gene status are assigned to Group I, while patients with deleted/mutant p53 gene status are assigned to Group II.

GROUP I: Starting with week 2, patients receive navtemadlin as in Step 1 and undergo radiation therapy (RT) daily for 5 weeks in the absence of disease progression or unacceptable toxicity, followed by surgery 5-8 weeks after RT completion.

GROUP II: Starting with week 2, patients undergo radiation therapy daily for 5 weeks in the absence of disease progression or unacceptable toxicity, followed by surgery 5-8 weeks after RT completion.

After completion of study treatment, patients are followed up every 3 months for 2 years, and then at 2.5 years.

ELIGIBILITY:
Inclusion Criteria:

* PRIOR TO STEP 1 REGISTRATION INCLUSION CRITERIA
* Patients with pathologically proven diagnosis of grade 2-3 (intermediate or high grade) soft tissue sarcoma with size >= 5 cm are eligible to enroll if the intention to treat is curative. They must have sufficient tissue to submit to central laboratory for review as well as for NGS sequencing (see submission requirement). Biopsy should be obtained within 180 days prior to registration. Availability of tumor tissue is mandatory for study eligibility. The patient must have consented to provide archived formalin-fixed paraffin-embedded tumor tissue for future central pathology review, NGS sequencing and/or translational research
* Appropriate stage for study entry based on the following diagnostic workup:

  * History/physical examination within 30 days prior to registration;
  * Imaging of the primary tumor by MRI and/or computed tomography (CT) with or without contrast and/or positron emission tomography (PET)/CT within 30 days prior to registration;
  * Staging workup evaluated by chest CT and/or PET/CT showing no distant metastasis within 30 days prior to registration
* There is a planned definitive surgical resection of the primary tumor
* Eastern Cooperative Oncology Group (ECOG) or Zubrod performance status of 0-1 within 30 days prior to registration
* Absolute neutrophil count >= 1500/uL (within 30 days prior to registration)
* Platelet count >= 100,000/uL (within 30 days prior to registration)
* Hemoglobin: >= 10 g/dL (transfuse as necessary to raise levels; no transfusions within 7 days of start) (within 30 days prior to registration)
* Calculated creatinine clearance >= 60 ml/min (by Cockcroft-Gault formula) within 30 days prior to registration
* The patient has an adequate coagulation function as defined by international normalized ratio (INR) =< 1.5 x upper limit of normal (ULN) or prothrombin time (PT) =< 1.5 x ULN, and partial thromboplastin time (PTT or aPTT) =< 1.5 x ULN (those receiving anticoagulation therapy except low molecular weight heparin are excluded) (within 30 days prior to registration)
* Total bilirubin =< 1.5 x upper limit of normal (ULN) appropriate for age (except for patients with Gilbert's syndrome, who must have a total bilirubin < 3 mg/dL) (within 30 days prior to registration)
* Serum glutamic-oxaloacetic transaminase (SGOT) aspartate aminotransferase (AST) or serum glutamate pyruvate transaminase (SGPT) alanine aminotransaminase (ALT) < 2.5 upper limit of normal (ULN) appropriate for age (within 30 days prior to registration)
* Females of child-bearing potential must have a negative serum pregnancy test within 7 days prior to registration; exceptions: females not of child-bearing potential due to surgical sterilization (at least 6 weeks following tubal ligation, hysterectomy, or surgical bilateral oophorectomy with or without hysterectomy) confirmed by medical history; or female after menopause

  * A "postmenopausal woman" is a woman meeting either of the following criteria:

    * Spontaneous amenorrhea for at least 12 months, not induced by a medical condition such as anorexia nervosa and not taking medications during the amenorrhea that induced the amenorrhea (for example, oral contraceptives, hormones, gonadotropin releasing hormone, antiestrogens, selective estrogen receptor modulators [SERMs], or chemotherapy)
    * Spontaneous amenorrhea for 6 to 12 months and a follicle-stimulating hormone (FSH) level > 40 mIU/mL
  * Females of child-bearing potential and males must agree to use highly effective contraceptive precautions during the trial and up to 12 months following the last dose of study treatment; a highly effective method of birth control is defined as one that results in a low failure rate (that is, < 1% per year) when used consistently and correctly, such as implants, injectables, combined oral contraceptives, some intrauterine contraceptive devices (IUDs), sexual abstinence, or a vasectomized partner
* The patient or a legally authorized representative must provide study-specific informed consent prior to study entry
* PRIOR TO STEP 2 REGISTRATION INCLUSION CRITERIA
* TP53 sequencing by NGS performed by central pathology lab

Exclusion Criteria:

* PRIOR TO STEP 1 REGISTRATION EXCLUSION CRITERIA
* Well-differentiated liposarcoma or other low grade STS; Kaposi sarcoma, bone sarcomas, cartilage sarcomas and gastrointestinal stromal tumor (GIST)
* Definitive clinical or radiologic evidence of metastatic disease; indeterminant lung nodules less than 8 mm are acceptable
* The patient has history of another primary malignancy, with the exception of

  * Curatively treated non-melanomatous skin cancer;
  * Curatively treated cervical carcinoma in situ;
  * Non-metastatic prostate cancer
  * Other primary non-hematologic malignancies or solid tumor treated with curative intent, no known active disease, and no treatment administered during the last 3 years prior to registration
* The patient has a serious cardiac condition, such as congestive heart failure; New York Heart Association class II/ III/IV heart disease; unstable angina pectoris, cardiac stenting within 6 months of enrollment; myocardial infarction within the last 3 months; valvulopathy that is severe, moderate, or deemed clinically significant; or arrhythmias that are symptomatic or require treatment
* Females who are pregnant or breastfeeding
* Prior systemic chemotherapy for the study cancer (sarcoma); note that prior chemotherapy for a different cancer is allowable; however, unresolved toxicities from prior anti-tumor therapy, defined as not having resolved to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 grade 0 or 1, or to levels dictated in the eligibility criteria with the exception of alopecia (grade 2 or 3 toxicities from prior anti-tumor therapy that are considered irreversible [defined as having been present and stable for > 6 months], such as ifosfamide-related proteinuria, may be allowed if they are not otherwise described in the exclusion criteria AND there is agreement to allow by both the investigator and sponsor)
* Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields
* Clinically significant bleeding within 4 weeks of screening, current use of warfarin, factor Xa inhibitors, and direct thrombin inhibitors unless these medications can be safely discontinued 14 days prior to AMG-232 (KRT-232) administration; Note: low molecular weight heparin and prophylactic low dose warfarin are permitted; PT/PTT must meet the inclusion criteria; subjects taking warfarin must have their INR followed closely
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to AMG 232 (KRT-232)
* All subjects must agree to stop the use of all herbal medicines (e.g., St. John's wort), and supplements, within the 10 days prior to receiving the first dose of AMG 232 (KRT-232), and during the protocol AMG 232 (KRT-232) treatment (weeks 1-5); subjects may renew the use of the above at week 6; standard adult multi-vitamin is allowed
* All subjects must agree to stop the use of any known CYP3A4 substrates with narrow therapeutic window (such as alfentanil, astemizole, cisapride, dihydroergotamine, pimozide, quinidine, sirolimus, or terfenadine; within the 14 days prior to receiving the first dose of AMG 232 (KRT-232) and during protocol AMG 232 (KRT-232) treatment (weeks 1-5); other medications (such as fentanyl and oxycodone) may be allowed per investigator's assessment/evaluation
* All subjects must agree to stop the use of any known CYP2C8 substrates with a narrow therapeutic window within the 14 days prior to receiving the first dose of AMG 232 (KRT-232) and during protocol AMG 232 (KRT-232) treatment (weeks 1-5)
* All subjects are required to submit a list of medications consumed within 14 days prior to receiving the first dose of AMG232 (KRT-232) and during the protocol AMG232 (KRT-232) treatment (weeks 1-5)
* Patients with gastrointestinal (GI) tract disease causing the inability to take oral medication, malabsorption syndrome, requirement for intravenous alimentation, prior surgical procedures affecting absorption, uncontrolled inflammatory GI disease (e.g., Crohn's disease, ulcerative colitis), therefore could affect the absorption of AMG 232 (KRT-232) at the discretion of treating physician
* Patients with active infection requiring intravenous (IV) antibiotics within 2 weeks of registration
* Patients with known positive hepatitis B surface antigen (HepBsAg) (indicative of chronic hepatitis B), positive hepatitis total core antibody with negative HBsAG (suggestive of occult hepatitis B), or detectable hepatitis C virus RNA by a polymerase-chain reaction (PCR) assay (indicative of active hepatitis C - screening is generally done by hepatitis C antibody (HepCAb), followed by hepatitis C virus RNA by PCR if HepCAb is positive)
* Patients known to be positive for human immunodeficiency virus (HIV) are NOT excluded from this study, but HIV-positive patients must have:

  * A stable regimen of highly active anti-retroviral therapy (HAART)
  * No requirement for concurrent antibiotics or antifungal agents for the prevention of opportunistic infections
  * A CD4 count above 250 cells/mcL and an undetectable HIV viral load on standard PCR-based test
  * HIV testing is not required
* Treatment with medications known to cause corrected QT (QTc) interval prolongation within 7 days of study day 1 is not permitted unless approved by the sponsor; use of ondansetron is permitted for treatment of nausea and vomiting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2018-06-20 (Actual); Primary Completion 2023-08-27 (Actual); Study Completion 2025-09-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Meng X Welliver, Principal Investigator — NRG Oncology
Locations (53):
- United States (53):
  - CTCA at Western Regional Medical Center, Goodyear, Arizona
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - University of Arizona Cancer Center-Orange Grove Campus, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - CTCA at Southeastern Regional Medical Center, Newnan, Georgia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Eastern Regional Medical Center, Philadelphia, Pennsylvania
  - UPMC-Shadyside Hospital, Pittsburgh, Pennsylvania
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Aurora Health Center-Fond du Lac, Fond du Lac, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

REFERENCES:
- [Derived] Vatner R, James CD, Sathiaseelan V, Bondra KM, Kalapurakal JA, Houghton PJ. Radiation therapy and molecular-targeted agents in preclinical testing for immunotherapy, brain tumors, and sarcomas: Opportunities and challenges. Pediatr Blood Cancer. 2021 May;68 Suppl 2:e28439. doi: 10.1002/pbc.28439. Epub 2020 Aug 22. PMID 32827353
- [Derived] Elzanowska J, Semira C, Costa-Silva B. DNA in extracellular vesicles: biological and clinical aspects. Mol Oncol. 2021 Jun;15(6):1701-1714. doi: 10.1002/1878-0261.12777. Epub 2020 Aug 19. PMID 32767659

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is a two-step study in which all participants start one week of treatment at Step 1 at the current dose escalation level while p53 status is determined, but Step 2 assigns the full/remaining course of treatment and determines the intended analysis population: participants with wild-type p53 (Group I) continue on navtemadlin for the purpose of the study analysis, while the rest of participants (Group II) discontinue navtemadlin and are not included in endpoint analyses.
Groups:
- Step 1 (Tumor Tissue Testing, Navtemadlin): Cohort A: Patients undergo tumor tissue testing for p53 gene status and receive navtemadlin PO on days 2-4 of week 1 in the absence of disease progression or unacceptable toxicity. Cohort A = Patients with extremity/body wall soft tissue sarcoma. Dose escalates separately within each cohort.
- Step 1 (Tumor Tissue Testing, Navtemadlin): Cohort B: Patients undergo tumor tissue testing for p53 gene status and receive navtemadlin PO on days 2-5 of week 1 in the absence of disease progression or unacceptable toxicity. Cohort A = Patients with abdomen/pelvis/retroperitoneum soft tissue sarcoma. Dose escalates separately within each cohort.
- Step 2: Group I (Navtemadlin, Radiation Therapy, Surgery): Starting with week 2, patients receive navtemadlin as in Step 1 and undergo radiation therapy (RT) daily for 5 weeks in the absence of disease progression or unacceptable toxicity, followed by surgery 5-8 weeks after RT completion. Group I = Wild-type p53 status determined by testing in Step 1. (Both cohorts)
- Step 2: Group II (Radiation Therapy, Surgery): Starting with week 2, patients undergo radiation therapy daily for 5 weeks in the absence of disease progression or unacceptable toxicity, followed by surgery 5-8 weeks after RT completion. Group II = Mutant or unknown p53 status determined by testing in Step 1. (Both cohorts.)
Period: Total Enrollment to Step 1
Arm/Group | Step 1 (Tumor Tissue Testing, Navtemadlin): Cohort A | Step 1 (Tumor Tissue Testing, Navtemadlin): Cohort B | Step 2: Group I (Navtemadlin, Radiation Therapy, Surgery) | Step 2: Group II (Radiation Therapy, Surgery)
Started | 27 | 12 | 0 | 0
Completed | 27 | 12 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Step 1: Dose Level 1
Arm/Group | Step 1 (Tumor Tissue Testing, Navtemadlin): Cohort A | Step 1 (Tumor Tissue Testing, Navtemadlin): Cohort B | Step 2: Group I (Navtemadlin, Radiation Therapy, Surgery) | Step 2: Group II (Radiation Therapy, Surgery)
Started | 4 | 5 | 0 | 0
Eligible | 4 | 5 | 0 | 0
Started Treatment | 3 | 5 | 0 | 0
Determined to Have Wild-type p53 (Group I) | 3 | 3 | 0 | 0
Determined to Have Mutant or Unknown p53 (Group II) | 0 | 2 | 0 | 0
Completed (Participants continuing to Step 2) | 3 | 5 | 0 | 0
Not Completed | 1 | 0 | 0 | 0
Not completed — Did not start protocol treatment | 1 | 0 | 0 | 0
Period: Step 1: Dose Level 2
Arm/Group | Step 1 (Tumor Tissue Testing, Navtemadlin): Cohort A | Step 1 (Tumor Tissue Testing, Navtemadlin): Cohort B | Step 2: Group I (Navtemadlin, Radiation Therapy, Surgery) | Step 2: Group II (Radiation Therapy, Surgery)
Started | 7 | 7 | 0 | 0
Eligible | 7 | 7 | 0 | 0
Started Treatment | 6 | 5 | 0 | 0
Determined to Have Wild-type p53 (Group I) | 4 | 3 | 0 | 0
Determined to Have Mutant or Unknown p53 (Group II) | 2 | 2 | 0 | 0
Completed | 6 | 5 | 0 | 0
Not Completed | 1 | 2 | 0 | 0
Not completed — Did not start protocol treatment | 1 | 2 | 0 | 0
Period: Step 1: Dose Level 3
Arm/Group | Step 1 (Tumor Tissue Testing, Navtemadlin): Cohort A | Step 1 (Tumor Tissue Testing, Navtemadlin): Cohort B | Step 2: Group I (Navtemadlin, Radiation Therapy, Surgery) | Step 2: Group II (Radiation Therapy, Surgery)
Started | 16 | 0 | 0 | 0
Eligible | 16 | 0 | 0 | 0
Started Treatment | 15 | 0 | 0 | 0
Determined to Have Wild-type p53 (Group I) | 9 | 0 | 0 | 0
Determined to Have Mutant or Unknown p53 (Group II) | 6 | 0 | 0 | 0
Completed | 15 | 0 | 0 | 0
Not Completed | 1 | 0 | 0 | 0
Not completed — Did not start treatment | 1 | 0 | 0 | 0
Period: Step 2
Arm/Group | Step 1 (Tumor Tissue Testing, Navtemadlin): Cohort A | Step 1 (Tumor Tissue Testing, Navtemadlin): Cohort B | Step 2: Group I (Navtemadlin, Radiation Therapy, Surgery) | Step 2: Group II (Radiation Therapy, Surgery)
Started | 0 | 0 | 22 | 12
AE Reporting | 0 | 0 | 22 | 12
Protocol Endpoint Reporting (Only Group I participants are included in study endpoint analysis per design) | 0 | 0 | 22 | 0
Completed (Participants contributing data to study endpoint results or AE reporting are considered to have completed the study.) | 0 | 0 | 22 | 12
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Eligible participants who started protocol treatment.
Groups:
- Group I: Cohort A: Dose Level 1 (3x/Week): Patients undergo tumor tissue testing for p53 gene status and receive navtemadlin PO on days 2-4 of week 1 in the absence of disease progression or unacceptable toxicity. (Step 1) Starting with week 2, patients receive navtemadlin as in Step 1 and undergo radiation therapy daily for 5 weeks in the absence of disease progression or unacceptable toxicity, followed by surgery 5-8 weeks after RT completion.
  Group I = wild-type p53 status. Cohort A = Patients with extremity/body wall soft tissue sarcoma.
- Group I: Dose Level 2 (4x/Week): Patients undergo tumor tissue testing for p53 gene status and receive navtemadlin PO on days 2-5 of week 1 in the absence of disease progression or unacceptable toxicity. (Step 1) Starting with week 2, patients receive navtemadlin as in Step 1 and undergo radiation therapy daily for 5 weeks in the absence of disease progression or unacceptable toxicity, followed by surgery 5-8 weeks after RT completion.
  Group I = wild-type p53 status. Cohort A = Patients with extremity/body wall soft tissue sarcoma.
- Group I: Cohort A: Dose Level 3 (5x/Week): Patients undergo tumor tissue testing for p53 gene status and receive navtemadlin PO on days 1-5 of week 1 in the absence of disease progression or unacceptable toxicity. (Step 1) Starting with week 2, patients receive navtemadlin as in Step 1 and undergo radiation therapy daily for 5 weeks in the absence of disease progression or unacceptable toxicity, followed by surgery 5-8 weeks after RT completion.
  Group I = wild-type p53 status. Cohort A = Patients with extremity/body wall soft tissue sarcoma.wall soft tissue sarcoma.
- Group I: Cohort B: Dose Level 1 (3x/Week): Patients undergo tumor tissue testing for p53 gene status and receive navtemadlin PO on days 2-4 of week 1 in the absence of disease progression or unacceptable toxicity. (Step 1) Starting with week 2, patients receive navtemadlin as in Step 1 and undergo radiation therapy daily for 5 weeks in the absence of disease progression or unacceptable toxicity, followed by surgery 5-8 weeks after RT completion.
  Group I = wild-type p53 status. Cohort B = Patients with abdomen/pelvis/retroperitoneum soft tissue sarcoma.
- Group I: Cohort B: Dose Level 2 (4x/Week): Patients undergo tumor tissue testing for p53 gene status and receive navtemadlin PO on days 2-5 of week 1 in the absence of disease progression or unacceptable toxicity. (Step 1) Starting with week 2, patients receive navtemadlin as in Step 1 and undergo radiation therapy daily for 5 weeks in the absence of disease progression or unacceptable toxicity, followed by surgery 5-8 weeks after RT completion.
  Group I = wild-type p53 status. Cohort B = Patients with abdomen/pelvis/retroperitoneum soft tissue sarcoma.
- Group II: Cohort A: Level 2 (4x/Week): Patients undergo tumor tissue testing for p53 gene status and receive navtemadlin PO on days 2-5 of week 1 in the absence of disease progression or unacceptable toxicity. Starting with week 2, patients undergo radiation therapy daily for 5 weeks in the absence of disease progression or unacceptable toxicity, followed by surgery 5-8 weeks after RT completion. Group II = mutant or unknown p53 status. Cohort A = Patients with extremity/body wall soft tissue sarcoma.
- Group II: Cohort A: Dose Level 3 (5x/Week): Patients undergo tumor tissue testing for p53 gene status and receive navtemadlin PO on days 1-5 of week 1 in the absence of disease progression or unacceptable toxicity. Starting with week 2, patients undergo radiation therapy daily for 5 weeks in the absence of disease progression or unacceptable toxicity, followed by surgery 5-8 weeks after RT completion. Group II = mutant or unknown p53 status. Cohort A = Patients with extremity/body wall soft tissue sarcoma.
- Group II: Cohort B: Dose Level 1 (3x/Week): Patients undergo tumor tissue testing for p53 gene status and receive navtemadlin PO on days 2-4 of week 1 in the absence of disease progression or unacceptable toxicity. Starting with week 2, patients undergo radiation therapy daily for 5 weeks in the absence of disease progression or unacceptable toxicity, followed by surgery 5-8 weeks after RT completion. Group II = mutant or unknown p53 status. Cohort B = Patients with abdomen/pelvis/retroperitoneum soft tissue sarcoma.
- Group II: Cohort B: Dose Level 2 (4x/Week): Patients undergo tumor tissue testing for p53 gene status and receive navtemadlin PO on days 2-5 of week 1 in the absence of disease progression or unacceptable toxicity. Starting with week 2, patients undergo radiation therapy daily for 5 weeks in the absence of disease progression or unacceptable toxicity, followed by surgery 5-8 weeks after RT completion. Group II = mutant or unknown p53 status. Cohort B = Patients with abdomen/pelvis/retroperitoneum soft tissue sarcoma.
- Total: Total of all reporting groups
Arm/Group | Group I: Cohort A: Dose Level 1 (3x/Week) | Group I: Dose Level 2 (4x/Week) | Group I: Cohort A: Dose Level 3 (5x/Week) | Group I: Cohort B: Dose Level 1 (3x/Week) | Group I: Cohort B: Dose Level 2 (4x/Week) | Group II: Cohort A: Level 2 (4x/Week) | Group II: Cohort A: Dose Level 3 (5x/Week) | Group II: Cohort B: Dose Level 1 (3x/Week) | Group II: Cohort B: Dose Level 2 (4x/Week) | Total
Number analyzed (Participants) | 3 | 4 | 9 | 3 | 3 | 2 | 6 | 2 | 2 | 34
Age, Customized [Count of Participants; unit: Participants]
  ≤ 49 years | 0 | 0 | 4 | 0 | 0 | 0 | 1 | 0 | 1 | 6
  50 - 59 years | 0 | 0 | 1 | 1 | 0 | 2 | 1 | 0 | 1 | 6
  60 -69 years | 3 | 4 | 1 | 2 | 2 | 0 | 3 | 1 | 0 | 16
  ≥ 70 years | 0 | 0 | 3 | 0 | 1 | 0 | 1 | 1 | 0 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 6 | 2 | 1 | 2 | 4 | 1 | 1 | 19
  Male | 2 | 3 | 3 | 1 | 2 | 0 | 2 | 1 | 1 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 3 | 4 | 8 | 2 | 3 | 2 | 5 | 2 | 2 | 31
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 6
  White | 3 | 2 | 7 | 3 | 0 | 2 | 5 | 2 | 1 | 25
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2
Zubrod performance status [Count of Participants; unit: Participants] — 0 = Asymptomatic; 1 = Symptomatic but completely ambulatory; 2 = Symptomatic, <50% in bed during the day; 3 = Symptomatic, >50% in bed, but not bedbound; 4 = Bedbound; 5 = Death
  Participants
    0 | 0 | 2 | 7 | 2 | 2 | 1 | 5 | 2 | 1 | 22
    1 | 3 | 2 | 2 | 1 | 1 | 1 | 1 | 0 | 1 | 12
Histology from Central Review [Count of Participants; unit: Participants] — A description of a tumor based on how the cancer cells and tissue look under a microscope. Population: One participant's tissue was not centrally reviewed.
  Participants
    number analyzed (Participants) | 3 | 4 | 9 | 3 | 3 | 2 | 5 | 2 | 2 | 33
    Dedifferentiated liposarcoma | 0 | 1 | 0 | 2 | 2 | 0 | 1 | 0 | 1 | 7
    Extraskeletal myxoid chondrosarcoma | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
    Malignant peripheral nerve sheath tumor | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
    Myxofibrosarcoma | 2 | 2 | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 8
    Myxoid liposarcoma | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
    Synovial sarcoma | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2
    Undifferentiated pleomorphic sarcoma | 0 | 0 | 2 | 0 | 0 | 1 | 4 | 0 | 0 | 7
    Undifferentiated spindle cell sarcoma | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
    Leiomyosarcoma | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
    Solitary fibrous tumor | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
    Liposarcoma, not otherwise specified | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 3
Histologic Grade from Central Review [Count of Participants; unit: Participants] — Sarcoma grade is determined using the Fédération Nationale des Centres de Lutte Contre le Cancer (FNCLCC) system, which is based and is based on 3 scored factors:
  * Differentiation: How the cancer cells look: 1 (a lot like normal cells) to 3 (very abnormal)
  * Mitotic count: How many cancer cells seen dividing: 1 (less) to 3 (more).
  * Tumor necrosis: How much of the tumor is made up of dying tissue: 0 (less) to 2 (more).
  The sum of the 3 scores determines the grade: 2,3 = Grade I; 4,5 = Grade II; 6,7,8 = Grade III. Lower grade indicates better prognosis. Population: One participant's tissue was not centrally reviewed.
  Participants
    number analyzed (Participants) | 3 | 4 | 9 | 3 | 3 | 2 | 5 | 2 | 2 | 33
    Grade II | 2 | 0 | 2 | 1 | 2 | 0 | 0 | 0 | 1 | 8
    Grade III | 1 | 4 | 7 | 2 | 1 | 2 | 5 | 2 | 1 | 25
Primary tumor site [Count of Participants; unit: Participants]
  Back | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Buttock | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2
  Distal Lower Extremity | 1 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 5
  Distal Upper Extremity | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Proximal Lower Extremity | 1 | 3 | 4 | 0 | 0 | 0 | 2 | 0 | 0 | 10
  Proximal Upper Extremity | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Abdomen | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2
  Retroperitoneum | 0 | 0 | 0 | 2 | 3 | 0 | 0 | 1 | 1 | 7
  Pelvis | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Shoulder | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 3
Tumor size (cm) [Count of Participants; unit: Participants]
  5 - < 10 cm | 2 | 3 | 2 | 0 | 1 | 0 | 3 | 0 | 1 | 12
  10 - < 15 cm | 0 | 1 | 4 | 2 | 1 | 1 | 3 | 2 | 0 | 14
  ≥ 15 cm | 1 | 0 | 3 | 1 | 1 | 1 | 0 | 0 | 1 | 8

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) / Recommended Phase 2 Dosage for Each Cohort
Description: Dose was determined separately for each cohort using the classic 3+3 design to determine the safety of each dose level from the number of participants with dose limiting toxicities (DLTs), starting with dose level 1. If dose level 1 were considered unsafe, a lower dose level of twice/week would be tested. The highest dose level deemed safe is considered the MTD. Five additional patients were accrued to the MTD to ensure safety.
  A DLT is defined as any grade 4-5 adverse event (AE) using the Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v5.0) that was definitely, probably, or possibly (DPP) related to navtemadlin or combined navtemadlin+RT ≤ 4 weeks after completing navtemadlin. Any grade 3 AE DPP related to navtemadlin/navtemadlin+RT was also considered a DLT if due to the grade 3 AE there was a delay of >2 weeks or if there were ≥ 2 dose reductions. CTCAE 5.0 Grade 3 is a severe AE, Grade 4 is a life-threatening or disabling AE, and Grade 5 results in death.
Time Frame: Baseline to end of navtemadlin + 4 weeks (approximately 10 weeks total)
Population: Eligible wild-type p53 participants who either received at least one dose of navtemadlin if there was a dose limiting toxicity (DLT), or, in the absence of DLT, received at least one fraction of RT and completed DLT observation period (4 weeks after completion of navtemadlin). Step 2 Group I participants (Group I = wild-type p53 status).
Measure: Number; unit: times per week of 125mg PO
Groups:
- Cohort A; Cohort B: All participants who received at least one dose of 120 mg navtemadlin PO either 3 times/week (Dose Level 1), 4 times/week (Dose Level 2), or 5 times/week (Dose Level 3). Planned dosing was for six weeks; 50 Gy RT over 5 weeks starting week 2 day 1; surgery 5-8 weeks after RT completion.
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 15 | 6
times per week of 125mg PO | 5 | NA — The study closed due to poor accrual during dose level 2 and therefore MTD could not be determined.

2. Primary Outcome: Number of Participants Who Experienced Dose-limiting Toxicities (DLTs)
Description: A DLT is defined as any grade 4-5 adverse event (AE) using the Common Terminology Criteria for Adverse Events Version 5.0 (CTCAE v5.0) that was definitely, probably, or possibly related to navtemadlin or combined navtemadlin+RT up to 4 weeks after the completion of navtemadlin. Any grade 3 AE definitely, probably, or possibly related to navtemadlin or combined navtemadlin+RT was also considered DLT if any of the 2 following situations occurred: a delay of >2 weeks due to the grade 3 AE, or ≥ 2 dose reductions due to the grade 3 AE. CTCAE 5.0 Grade 3 is a severe AE, Grade 4 is a life-threatening or disabling AE, and Grade 5 results in death.
Time Frame: Baseline to end of navtemadlin + 4 weeks (approximately 10 weeks total)
Population: Eligible wild-type p53 participants who either received at least one dose of navtemadlin if there was a dose limiting toxicity (DLT), or, in the absence of DLT, received at least one fraction of RT and completed DLT observation period (4 weeks after completion of navtemadlin).
Measure: Count of Participants; unit: Participants
Groups:
- Cohort A: Dose Level 1 (3x/Week): Step 1: Patients undergo tumor tissue testing for p53 gene status and receive navtemadlin PO on days 2-4 of week 1 in the absence of disease progression or unacceptable toxicity.
  Step 2: Starting with week 2, patients receive navtemadlin as in Step 1 and undergo radiation therapy daily for 5 weeks in the absence of disease progression or unacceptable toxicity, followed by surgery 5-8 weeks after RT completion.
  Cohort A = Patients with extremity/body wall soft tissue sarcoma.
- Cohort A: Dose Level 2 (4x/Week): Step 1: Patients undergo tumor tissue testing for p53 gene status and receive navtemadlin PO on days 2-5 of week 1 in the absence of disease progression or unacceptable toxicity.
  Step 2: Starting with week 2, patients receive navtemadlin as in Step 1 and undergo radiation therapy daily for 5 weeks in the absence of disease progression or unacceptable toxicity, followed by surgery 5-8 weeks after RT completion.
  Cohort A = Patients with extremity/body wall soft tissue sarcoma.
- Cohort A: Dose Level 3 (5x/Week): Step 1: Patients undergo tumor tissue testing for p53 gene status and receive navtemadlin PO on days 1-5 of week 1 in the absence of disease progression or unacceptable toxicity.
  Step 2: Starting with week 2, patients receive navtemadlin as in Step 1 and undergo radiation therapy daily for 5 weeks in the absence of disease progression or unacceptable toxicity, followed by surgery 5-8 weeks after RT completion.
  Cohort A = Patients with extremity/body wall soft tissue sarcoma.wall soft tissue sarcoma.
- Cohort B: Dose Level 1 (3x/Week): Step 1: Patients undergo tumor tissue testing for p53 gene status and receive navtemadlin PO on days 2-4 of week 1 in the absence of disease progression or unacceptable toxicity.
  Step 2: Starting with week 2, patients receive navtemadlin as in Step 1 and undergo radiation therapy daily for 5 weeks in the absence of disease progression or unacceptable toxicity, followed by surgery 5-8 weeks after RT completion.
  Cohort B = Patients with abdomen/pelvis/retroperitoneum soft tissue sarcoma.
- Cohort B: Dose Level 2 (4x/Week): Step 1: Patients undergo tumor tissue testing for p53 gene status and receive navtemadlin PO on days 2-5 of week 1 in the absence of disease progression or unacceptable toxicity.
  Step 2: Starting with week 2, patients receive navtemadlin as in Step 1 and undergo radiation therapy daily for 5 weeks in the absence of disease progression or unacceptable toxicity, followed by surgery 5-8 weeks after RT completion.
  Cohort B = Patients with abdomen/pelvis/retroperitoneum soft tissue sarcoma.
Arm/Group | Cohort A: Dose Level 1 (3x/Week) | Cohort A: Dose Level 2 (4x/Week) | Cohort A: Dose Level 3 (5x/Week) | Cohort B: Dose Level 1 (3x/Week) | Cohort B: Dose Level 2 (4x/Week)
Number analyzed (Participants) | 3 | 4 | 8 | 3 | 3
Participants | 0 | 0 | 0 | 0 | 1

3. Secondary Outcome: Percent of Necrosis in Final Surgical Resection Specimen
Description: The evaluation for pathologic response will include a formal evaluation of percent necrosis according to the guidelines established for osteosarcoma and is determined by central pathological review.
Time Frame: At time of surgery (approximately 11 to 14 weeks)
Population: Eligible Group I (wild-type p53) participants who started protocol treatment and had central pathological review of their final surgical resection specimen.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Dose Level 1 (3x/Week) | Cohort A: Dose Level 2 (4x/Week) | Cohort A: Dose Level 3 (5x/Week) | Cohort B: Dose Level 1 (3x/Week) | Cohort B: Dose Level 2 (4x/Week)
Number analyzed (Participants) | 3 | 2 | 8 | 3 | 1
Participants
  76-99% | 0 | 0 | 2 | 0 | 0
  50-75% | 0 | 0 | 2 | 0 | 0
  25-49% | 1 | 2 | 1 | 1 | 0
  <25% | 2 | 0 | 3 | 2 | 1

4. Secondary Outcome: Number of Participants With Pathologic Complete Response (PCR) in Final Surgical Resection Specimen
Description: Pathologic complete response is defined as 100% necrosis and is determined by central pathology review.
Time Frame: At time of surgery (approximately 11 to 14 weeks)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Groups:
- Cohort A: Dose Level 3 (5x/Week): Step 1: Patients undergo tumor tissue testing for p53 gene status and receive navtemadlin PO on days 1-5 of week 1 in the absence of disease progression or unacceptable toxicity.
  Step 2: Starting with week 2, patients receive navtemadlin as in Step 1 and undergo radiation therapy daily for 5 weeks in the absence of disease progression or unacceptable toxicity, followed by surgery 5-8 weeks after RT completion.
  Cohort A = Patients with extremity/body wall soft tissue sarcoma.
Arm/Group | Cohort A: Dose Level 1 (3x/Week) | Cohort A: Dose Level 2 (4x/Week) | Cohort A: Dose Level 3 (5x/Week) | Cohort B: Dose Level 1 (3x/Week) | Cohort B: Dose Level 2 (4x/Week)
Number analyzed (Participants) | 3 | 2 | 8 | 3 | 1
Participants | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Number of Participants With Local Failure
Description: Local failure (LF) was defined as local recurrence or progression after surgery, or amputation for treatment complications or recurrence/progression. In addition, any patient that did not have surgery was considered to have local failure. Local progression was defined as at lease 20% increase in the maximal dimension of the primary tumor taking as reference the smallest maximal dimension recorded since treatment started.
Time Frame: Baseline to the date of failure or last known follow-up, up to 2.5 years from end of RT (six weeks).
Population: Eligible Group I (wild-type p53) participants who started protocol treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort A: Dose Level 2 (4x/Week): Step 1: Patients undergo tumor tissue testing for p53 gene status and receive navtemadlin PO on days 2-4 of week 1 in the absence of disease progression or unacceptable toxicity.
  Step 2: Starting with week 2, patients receive navtemadlin as in Step 1 and undergo radiation therapy daily for 5 weeks in the absence of disease progression or unacceptable toxicity, followed by surgery 5-8 weeks after RT completion.
  Cohort A = Patients with extremity/body wall soft tissue sarcoma.
Arm/Group | Cohort A: Dose Level 1 (3x/Week) | Cohort A: Dose Level 2 (4x/Week) | Cohort A: Dose Level 3 (5x/Week) | Cohort B: Dose Level 1 (3x/Week) | Cohort B: Dose Level 2 (4x/Week)
Number analyzed (Participants) | 3 | 4 | 9 | 3 | 3
Participants | 1 | 2 | 2 | 1 | 1

6. Secondary Outcome: Number of Participants With Disease or Death From Any Cause
Description: Disease is defined as any of the following:
  Local, regional, or distant disease.
  * Local disease: tumor recurrence or progression. Progression is defined as at 20% increase in the maximal dimension of the primary tumor taking as reference the smallest maximal dimension recorded since treatment started;
  * Regional disease: Any nodal metastasis adjacent to the primary soft tissue sarcoma;
  * Distant disease: Any tumor that develops distantly from the primary site of sarcoma;
  * Amputation for treatment complications or recurrence/progression.
  * Failure to continue to surgery.
Time Frame: Baseline to the date of disease, death, or last known follow-up, up to 2.5 years from end of RT (six weeks).
Population: Eligible Group I (wild-type p53) participants who started protocol treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort A: Dose Level 3 (5x/Week): Step 1: Patients undergo tumor tissue testing for p53 gene status and receive navtemadlin PO on days 2-5 of week 1 in the absence of disease progression or unacceptable toxicity.
  Step 2: Starting with week 2, patients receive navtemadlin as in Step 1 and undergo radiation therapy daily for 5 weeks in the absence of disease progression or unacceptable toxicity, followed by surgery 5-8 weeks after RT completion.
  Cohort A = Patients with extremity/body wall soft tissue sarcoma.
- Cohort B: Dose Level 2 (4x/Week): Step 1: Patients undergo tumor tissue testing for p53 gene status and receive navtemadlin PO on days 2-4 of week 1 in the absence of disease progression or unacceptable toxicity.
  Step 2: Starting with week 2, patients receive navtemadlin as in Step 1 and undergo radiation therapy daily for 5 weeks in the absence of disease progression or unacceptable toxicity, followed by surgery 5-8 weeks after RT completion.
  Cohort B = Patients with abdomen/pelvis/retroperitoneum soft tissue sarcoma.
Arm/Group | Cohort A: Dose Level 1 (3x/Week) | Cohort A: Dose Level 2 (4x/Week) | Cohort A: Dose Level 3 (5x/Week) | Cohort B: Dose Level 1 (3x/Week) | Cohort B: Dose Level 2 (4x/Week)
Number analyzed (Participants) | 3 | 4 | 9 | 3 | 3
Participants | 1 | 2 | 4 | 1 | 1

7. Secondary Outcome: Number of Participants Who Died
Description: Death from any cause
Time Frame: Baseline to the date of death or last known follow-up, up to 2.5 years from end of RT (six weeks).
Population: Eligible Group I (wild-type p53) participants who started protocol treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort A: Dose Level 3 (5x/Week): Step 1: Patients undergo tumor tissue testing for p53 gene status and receive navtemadlin PO on days 1-5 of week 1 in the absence of disease progression or unacceptable toxicity.
  Step 2: Starting with week 2, patients receive navtemadlin as in Step 1 and undergo radiation therapy daily for 5 weeks in the absence of disease progression or unacceptable toxicity, followed by surgery 5-8 weeks after RT completion.
  Cohort A = Patients with extremity/body wall soft tissue sarcoma.
  .
Arm/Group | Cohort A: Dose Level 1 (3x/Week) | Cohort A: Dose Level 2 (4x/Week) | Cohort A: Dose Level 3 (5x/Week) | Cohort B: Dose Level 1 (3x/Week) | Cohort B: Dose Level 2 (4x/Week)
Number analyzed (Participants) | 3 | 4 | 9 | 3 | 3
Participants | 0 | 1 | 1 | 1 | 1

8. Secondary Outcome: Serial Serum Macrophage Inhibitory Cytokine-1 Levels
Description: Will be tabulated and descriptive statistics and calculated for each dose level.
Time Frame: Up to 2.5 years
Reporting Status: Not Posted, anticipated posting 2026-06

9. Secondary Outcome: Navtemadlin Exposure-response Relationships
Time Frame: Up to 2.5 years
Reporting Status: Not Posted, anticipated posting 2026-06

10. Other Pre Specified Outcome: Tumor Volume Changes
Description: Will be compared by paired t test.
Time Frame: Up to 2.5 years
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Clinical Outcomes by Genomic Biomarkers
Time Frame: Up to 2.5 years
Reporting Status: Not Posted

12. Other Pre Specified Outcome: mdm2/4 Expression
Description: Will be correlated with protein levels and assessed using Pearson's correlation.
Time Frame: Up to 2.5 years
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Tumor Genetic Mutations in Deoxyribonucleic Acid Ribonucleic Acid Isolated From Exosomes
Time Frame: Up to 2.5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Baseline to 2.5 years from end of RT (six weeks).
Groups:
- Group I: Cohort A: Dose Level 1 (3x/Week): Step 1: Patients undergo tumor tissue testing for p53 gene status and receive navtemadlin PO on days 2-4 of week 1 in the absence of disease progression or unacceptable toxicity.
  Step 2: Starting with week 2, patients receive navtemadlin as in Step 1 and undergo radiation therapy daily for 5 weeks in the absence of disease progression or unacceptable toxicity, followed by surgery 5-8 weeks after RT completion.
  Group I = Wild-type p53. Cohort A = Patients with extremity/body wall soft tissue sarcoma.
- Group I: Cohort A: Dose Level 2 (4x/Week): Step 1: Patients undergo tumor tissue testing for p53 gene status and receive navtemadlin PO on days 2-5 of week 1 in the absence of disease progression or unacceptable toxicity.
  Step 2: Starting with week 2, patients receive navtemadlin as in Step 1 and undergo radiation therapy daily for 5 weeks in the absence of disease progression or unacceptable toxicity, followed by surgery 5-8 weeks after RT completion.
  Group I = Wild-type p53. Cohort A = Patients with extremity/body wall soft tissue sarcoma.
- Group I: Cohort A: Dose Level 3 (5x/Week): Step 1: Patients undergo tumor tissue testing for p53 gene status and receive navtemadlin PO on days 1-5 of week 1 in the absence of disease progression or unacceptable toxicity.
  Step 2: Starting with week 2, patients receive navtemadlin as in Step 1 and undergo radiation therapy daily for 5 weeks in the absence of disease progression or unacceptable toxicity, followed by surgery 5-8 weeks after RT completion.
  Group I = Wild-type p53. Cohort A = Patients with extremity/body wall soft tissue sarcoma.
- Group I: Cohort B: Dose Level 1 (3x/Week); Group I: Cohort B: Dose Level 2 (4x/Week): Step 1: Patients undergo tumor tissue testing for p53 gene status and receive navtemadlin PO on days 2-4 of week 1 in the absence of disease progression or unacceptable toxicity.
  Step 2: Starting with week 2, patients receive navtemadlin as in Step 1 and undergo radiation therapy daily for 5 weeks in the absence of disease progression or unacceptable toxicity, followed by surgery 5-8 weeks after RT completion.
  Group I = Wild-type p53. Cohort B = Patients with abdomen/pelvis/retroperitoneum soft tissue sarcoma.
- Group II: Cohort A: Dose Level 2 (4x/Week): Step 1: Patients undergo tumor tissue testing for p53 gene status and receive navtemadlin PO on days 2-4 of week 1 in the absence of disease progression or unacceptable toxicity.
  Step 2: Starting with week 2, patients undergo radiation therapy daily for 5 weeks in the absence of disease progression or unacceptable toxicity, followed by surgery 5-8 weeks after RT completion.
  Group II = Mutant/unknown p53. Cohort A = Patients with extremity/body wall soft tissue sarcoma.
- Group II: Cohort A: Dose Level 3 (5x/Week): Step 1: Patients undergo tumor tissue testing for p53 gene status and receive navtemadlin PO on days 2-5 of week 1 in the absence of disease progression or unacceptable toxicity.
  Step 2: Starting with week 2, patients undergo radiation therapy daily for 5 weeks in the absence of disease progression or unacceptable toxicity, followed by surgery 5-8 weeks after RT completion.
  Group II = Mutant/unknown p53. Cohort A = Patients with extremity/body wall soft tissue sarcoma.
- Group II: Cohort B: Dose Level 1 (3x/Week); Group II: Cohort B: Dose Level 2 (4x/Week): Step 1: Patients undergo tumor tissue testing for p53 gene status and receive navtemadlin PO on days 2-4 of week 1 in the absence of disease progression or unacceptable toxicity.
  Step 2: Starting with week 2, patients undergo radiation therapy daily for 5 weeks in the absence of disease progression or unacceptable toxicity, followed by surgery 5-8 weeks after RT completion.
  Group II = Mutant/unknown p53. Cohort B = Patients with abdomen/pelvis/retroperitoneum soft tissue sarcoma.
Arm/Group | Group I: Cohort A: Dose Level 1 (3x/Week) | Group I: Cohort A: Dose Level 2 (4x/Week) | Group I: Cohort A: Dose Level 3 (5x/Week) | Group I: Cohort B: Dose Level 1 (3x/Week) | Group I: Cohort B: Dose Level 2 (4x/Week) | Group II: Cohort A: Dose Level 2 (4x/Week) | Group II: Cohort A: Dose Level 3 (5x/Week) | Group II: Cohort B: Dose Level 1 (3x/Week) | Group II: Cohort B: Dose Level 2 (4x/Week)
All-Cause Mortality (participants affected / at risk) | 0/3 | 1/4 | 1/9 | 1/3 | 1/3 | 1/2 | 0/6 | 1/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 2/3 | 4/4 | 5/9 | 3/3 | 3/3 | 1/2 | 1/6 | 1/2 | 1/2
Other Adverse Events (participants affected / at risk) | 3/3 | 4/4 | 9/9 | 3/3 | 3/3 | 2/2 | 6/6 | 2/2 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group I: Cohort A: Dose Level 1 (3x/Week) (N=3) | Group I: Cohort A: Dose Level 2 (4x/Week) (N=4) | Group I: Cohort A: Dose Level 3 (5x/Week) (N=9) | Group I: Cohort B: Dose Level 1 (3x/Week) (N=3) | Group I: Cohort B: Dose Level 2 (4x/Week) (N=3) | Group II: Cohort A: Dose Level 2 (4x/Week) (N=2) | Group II: Cohort A: Dose Level 3 (5x/Week) (N=6) | Group II: Cohort B: Dose Level 1 (3x/Week) (N=2) | Group II: Cohort B: Dose Level 2 (4x/Week) (N=2)
Anemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 1 | 3 | 0 | 1 | 0 | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Allergic reaction (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Viremia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seroma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Serum amylase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group I: Cohort A: Dose Level 1 (3x/Week) (N=3) | Group I: Cohort A: Dose Level 2 (4x/Week) (N=4) | Group I: Cohort A: Dose Level 3 (5x/Week) (N=9) | Group I: Cohort B: Dose Level 1 (3x/Week) (N=3) | Group I: Cohort B: Dose Level 2 (4x/Week) (N=3) | Group II: Cohort A: Dose Level 2 (4x/Week) (N=2) | Group II: Cohort A: Dose Level 3 (5x/Week) (N=6) | Group II: Cohort B: Dose Level 1 (3x/Week) (N=2) | Group II: Cohort B: Dose Level 2 (4x/Week) (N=2)
Anemia (Blood and lymphatic system disorders) | 3 | 0 | 3 | 1 | 0 | 1 | 2 | 1 | 1
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cardiac disorders - Other (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 0
Belching (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bloating (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 0 | 6 | 0 | 1 | 0 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 3 | 3 | 8 | 3 | 3 | 1 | 4 | 2 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 4 | 8 | 3 | 3 | 2 | 4 | 2 | 2
Oral dysesthesia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2 | 4 | 3 | 3 | 1 | 2 | 2 | 1
Chills (General disorders) | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Edema limbs (General disorders) | 0 | 0 | 5 | 0 | 0 | 0 | 1 | 0 | 0
Edema trunk (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 3 | 3 | 8 | 2 | 3 | 1 | 4 | 0 | 0
Fever (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 0
General disorders and administration site conditions - Other (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Localized edema (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pain (General disorders) | 2 | 1 | 2 | 0 | 1 | 1 | 1 | 0 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Infections and infestations - Other (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Papulopustular rash (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Thrush (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Viremia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Burn (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis radiation (Injury, poisoning and procedural complications) | 2 | 0 | 6 | 1 | 0 | 0 | 2 | 0 | 0
Injury, poisoning and procedural complications - Other (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Seroma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Alkaline phosphatase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Creatinine increased (Investigations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1
INR increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1
Investigations - Other (Investigations) | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 1 | 1 | 2 | 0 | 0 | 1 | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Serum amylase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Weight loss (Investigations) | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 4 | 7 | 2 | 1 | 1 | 1 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 4 | 0 | 0 | 0 | 2 | 0 | 0
Superficial soft tissue fibrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 2 | 3 | 0 | 1 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Muscle weakness left-sided (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nervous system disorders - Other (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paresthesia (Nervous system disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0
Confusion (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Renal and urinary disorders - Other (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary frequency (Renal and urinary disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary urgency (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 1 | 1 | 1 | 1 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Skin atrophy (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Skin induration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Thromboembolic event (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Dose escalates independently in each cohort (extremity/body wall; abdomen/pelvis/retroperitoneum). All participants begin one week of treatment at Step 1 while p53 determination takes place. At Step 2, participants with wild-type p53 continue study drug for purpose of study analysis. The rest discontinue study drug and are not included in study analysis; only collected AEs are reported. Study accrual stopped early due to poor accrual, therefore the third dose level did not open for Cohort B.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-01): https://cdn.clinicaltrials.gov/large-docs/66/NCT03217266/Prot_SAP_000.pdf